CLINICAL TRIAL: NCT01537588
Title: Changes in Muscle Morphology Resulting From ACL Reconstruction: Impact on Strength and Function
Brief Title: Changes in Muscle Morphology Resulting From Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: April 2009
Record Dates: First submitted 2012-02-14; First posted 2012-02-23 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Isolated Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament; hamstring; semitendinosus; gracilis; graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard (Active Comparator): ACL reconstruction with autograft harvest of STG from ACL-deficient leg
  Interventions: Other: Autograft STG harvest from ACL-deficient leg
- Autograft harvest of STG from ACL-deficient leg (Experimental): Autograft harvest of STG from leg contralateral to ACL-deficient leg
  Interventions: Other: Autograft harvest contralateral to ACL-deficient leg
- Normal matched (No Intervention)

INTERVENTIONS:
Other: Autograft STG harvest from ACL-deficient leg — Semitendinosus-gracilis graft harvest is undertaken on same limb that is undergoing ACL reconstruction
  Arms: Standard
Other: Autograft harvest contralateral to ACL-deficient leg — Semitendinosus-gracilis graft harvest is undertaken on limb contralateral to that undergoing ACL reconstruction
  Arms: Autograft harvest of STG from ACL-deficient leg

SUMMARY:
The aim of this study is to gain new knowledge on the impact of hamstring tendon harvest and apply that knowledge to the treatment and management of patients who undergo anterior cruciate ligament (ACL) reconstruction. There are three main components of this study:

1. How do muscle shape, size, strength, and ability to function change following hamstring grafting for ACL reconstruction;
2. How does physical activity change following ACL reconstruction;
3. Is there a difference in outcome if graft harvest is done from the injured versus uninjured limbs

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 50 years old; isolated ACL rupture confirmed on MRI

Exclusion Criteria:

* other physical or mental health issues that affect ability to complete rehabilitation and/or study follow-ups

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Muscle cross sectional area | 12 months post-surgery
  Measured on bilateral MRI taken from ischial tuberosity to 10 cm below knee joint line

SECONDARY OUTCOMES:
Knee flexion and extension isokinetic strength | 12-months post-surgery
  Eccentric anc concentric strength measured at 60, 150, and 270 degrees/second on dynamometer in sitting and in 5 degrees hip flexion
Physical activity | 12 months post-surgery
  7-day record of activity using accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila McRae, MSc, Principal Investigator — University of Manitoba, Pan Am Clinic Foundation
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada